CLINICAL TRIAL: NCT06795139
Title: Feasibility Pilot of a Trial Enrollment Diversity Dashboard (TEDD)
Brief Title: Pilot of a Trial Enrollment Diversity Dashboard
Acronym: TEDD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Society of Clinical Oncology (Other)
Responsible Party: Principal Investigator, Andrew Hantel, MD, Principle Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-544; K08CA273043-01 (NIH)
Record Dates: First submitted 2025-01-22; First posted 2025-01-27 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Leukemia; Acute Leukemia
Keywords: Leukemia; Acute Leukemia; Clinical Trial Diversity
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TEDD Intervention (Experimental): 12 medical professional participants will complete the following:
  * Baseline survey.
  * Usage and access of the TEDD intervention over a 12-month period.
  * Follow up surveys at the end of each quarter.
  Interventions: Behavioral: Trial Enrollment Diversity Dashboard Behavioral

INTERVENTIONS:
Behavioral: Trial Enrollment Diversity Dashboard Behavioral — A data management and classification algorithm tool that provides personalized enrollment diversity performance data for clinician review and which aims to overcome race-ethnic disparities in Leukemia clinical trial participation. Data inputs and the Dashboard are within existing HIPAA-complaint electronic health records systems used at Dana-Farber Cancer Institute, and utilization data metrics are collected through the Tableau software supporting the intervention.

SUMMARY:
The goal of this study is to test the feasibility of a data visualization tool called the Trial Enrollment Diversity Dashboard (TEDD) to ensure participant diversity in acute leukemia trial enrollment.

DETAILED DESCRIPTION:
This study is about testing a tool called the Trial Enrollment Diversity Dashboard (TEDD) to see if it can help increase diversity in cancer clinical trials, specifically for leukemia. Clinical trials are important for developing new cancer treatments, but not all groups are equally represented in these trials. This can lead to treatments that may not work as well for everyone.

The TEDD tool is designed to give medical professionals feedback on how diverse their patient enrollments are clinical trials. By using this tool, medical professionals can see if they are enrolling a diverse group of patients and make changes if needed.

The study will involve a small group of medical professionals who treat leukemia patients. They will use the TEDD tool and provide feedback on its usability and effectiveness. Study procedures include completion of surveys and usage of the TEDD intervention dashboard.

It is expected that about 12 medical professionals will take part in this research study. Participation in this research study is expected to last about 14 months.

The National Cancer Institute is providing funding for this research study.

ELIGIBILITY:
Inclusion Criteria Medical Professionals:

* Physician, nurse practitioner, or physician assistant

  -≥10% clinical effort (or one ½ day of clinic per week for those working <1 FTE)
* Treats adult patients with leukemia or related diseases at the study sites
* Ability to understand and willingness to provide informed consent
* Age 18 or older

Inclusion Criteria Participant Population:

* Age ≥18 years old
* Diagnosis of leukemia, lymphoma, myeloma, or related diseases
* Seen by a physician for this diagnosis at one of the study sites

Exclusion Criteria Medical Professionals:

-Listed member of the research team

Exclusion Criteria Participant Population:

-Participants without the diagnoses of interest listed above, participants not seen at the study sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
TEDD Utilization Rate | 12 months
  Utilization will be measured as the proportion of quarters where a participant accessed the dashboard divided by the total number of study quarters. Based on 12 participants over 4 three-month quarters, there are a total of 48 person-quarters available for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hantel, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu